CLINICAL TRIAL: NCT06410131
Title: A Phase 1, First-in-Human, Open-Label, Dose Escalation and Dose Expansion Study of FTL008.16, a Recombinant Anti-CD137 and Anti-5T4 Bispecific Antibody, in Patients With Advanced or Metastatic Solid Tumors
Brief Title: Study in Patients With Advanced Solid Tumors to Evaluate the Safety of FTL008.16
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sound Biopharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FTL008.16-101
Record Dates: First submitted 2024-04-30; First posted 2024-05-10 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumors
Keywords: Solid Tumors; Sound Biopharmaceuticals; FTL008.16

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 Part 1 Dose Escalation (Experimental): Escalating doses of FTL008.16 depending on cohort at enrollment
  Interventions: Drug: FTL008.16
- Arm 1 Part 2 Dose Expansion (Experimental): Two dose groups of FTL008.16 depending on data of Arm 1 Part 1
  Interventions: Drug: FTL008.16

INTERVENTIONS:
Drug: FTL008.16 — IV infusion every 2 weeks

SUMMARY:
This is an open, multi-center, multi-cohort phase I clinical study designed to evaluate safety, tolerability, pharmacokinetics and initial efficacy of FTL008.16 in patients with advanced and metastatic solid tumors.

DETAILED DESCRIPTION:
This study is divided into two phases: Part 1(dose escalation of FTL008.16) and Part 2(dose extension of FTL008.16), which is intended to include about 40 to 68 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the experiment and sign a written informed consent, with good compliance, and can follow the protocol visit plan and other research procedures.
2. Age ≥18 years and ≤75 years at the time of signing the informed consent, both male and female.
3. Expected survival ≥ 3 months.
4. Histologically or cytologically confirmed advanced solid tumors; The enrollment should focus on subjects with multiple solid tumor types/histologies likely to express 5T4 antigen, including but not limited to non-small cell lung cancer (NSCLC), stomach cancer, esophageal cancer, colorectal cancer, pancreatic cancer, head cancer, cervical squamous cell carcinoma, renal cell carcinoma, urothelial carcinoma, prostate cancer, breast cancer, ovary cancer, cervical cancer, endometrial cancer or malignant pleural mesothelioma.
5. Patients with advanced recurrence and metastasis of solid tumors with disease progression after standard treatment or intolerance to standard treatment or no standard treatment (definitions of standard treatment and recurrence refer to the latest CSCO guidelines or other authoritative diagnosis and treatment guidelines at home and abroad).
6. According to RECIST 1.1 solid tumor efficacy evaluation criteria, the patient had at least one lesion that could be measured or evaluated on imaging (CT, MRT); Patients enrolled in the extended study should have at least one measurable lesion; (Note: Tumor lesions that have previously received local treatment (such as radiotherapy, ablation, vascular intervention, etc.) will not be considered measurable unless there is sufficient evidence to demonstrate clear imaging progression of the lesion after local treatment).
7. Eastern Cancer Collaboration (ECOG) Physical fitness score of 0 or 1.
8. The patient must provide the required tumor tissue specimen (fresh tumor tissue or archived tumor tissue specimen).
9. The results of laboratory examination during the screening period indicate that the subject has good organ function;
10. If sexually active: females of childbearing potential must practice a medically effective methods of contraception during study participation and for at least 6 months after last dose of study drug.
11. If sexually active: men who are sexually active with females of child-bearing potential must agree to use highly effective methods of contraception during study participation and for at least 6 months after the last dose of study drug..

Exclusion Criteria:

1. History of hypersensitivity or idiosyncrasy to the excipients of the study drug or to any monoclonal antibody.
2. A history of malignancies other than the disease under study within the previous 5 years, with the exception of malignancies that have been cured after treatment and have no risk of recurrence (including but not limited to adequately treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell skin cancer, or breast ductal carcinoma in situ treated with radical surgery).
3. Systematic treatment with anti-tumor drugs (including chemotherapy, targeted therapy, antibody therapy, immunotherapy, endocrine therapy, etc.) was received within 4 weeks before the initial study.
4. Patients who have previously received cell immunotherapy (CAR-T).
5. Prior treatment with any anti-CD137/anti-5T4 antibody or drug (single agent or combination).
6. Adverse reactions caused by previous treatment did not recover to CTCAE (version 5.0) grade 1 or below (Alopecia, neurotoxicity returned to grade 2 or below, adverse reactions that the investigators judged were not a safety risk could be included);
7. Previously received allogeneic hematopoietic stem cell transplantation or solid organ transplantation;
8. Active primary or metastatic tumors of the central nervous system (except in patients who have previously been treated and have discontinued treatment 4 weeks prior to the first study drug administration, symptomless patients who do not require long-term glucocorticoid therapy), seizures, spinal cord compression, meningeal metastases, or carcinomatous meningitis.
9. Have or have suspected active autoimmune diseases, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, etc., but the following conditions can be included: Type 1 diabetes that can be controlled by alternative therapy alone, skin diseases that do not require systemic treatment (e.g. Psoriasis, vitiligo).
10. Suffering from pleural effusion, ascites or pericardial effusion that cannot be controlled by clinical symptoms or treatment.
11. Severe cardiovascular and cerebrovascular diseases, such as resting QTc interval ≥470ms (corrected QT interval, according to the Fridericia formula); Uncontrolled or poorly controlled hypertension (systolic more than 160mmHg or diastolic more than 100mmHg) or pulmonary hypertension; Unstable angina pectoris or myocardial infarction, coronary artery bypass grafting or stenting within 6 months prior to study administration; Chronic heart failure with heart function ≥2 (NYHA rating); Degree II and above heart block; Left ventricular ejection fraction (LVEF) less than 50%; Study cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months prior to medication.
12. History of pulmonary disease: interstitial pneumonia, obstructive pulmonary disease (requiring steroid treatment with a prednisone equivalent dose of more than 10mg/ day) or symptomatic bronchospasm.
13. Active tuberculosis (TB) is known to exist. Subjects suspected of active TB should be examined for chest X-rays, sputum, and clinical signs and symptoms.
14. An active infection requiring intravenous anti-infective treatment, or severe unhealed wounds or ulcers, occurs within 14 days prior to the first dose.
15. Positive human immunodeficiency virus (HIV) antibody test result, or active syphilis infection (i.e., positive treponema pallidum antibody and non-treponema pallidum antibody titer test result).
16. Autoimmune liver disease and decompensated cirrhosis; People with active hepatitis B virus or hepatitis C virus.
17. Systemic immunosuppressive therapy is required if received within 14 days before the first dose or during the trial. However, the following conditions were allowed: in the absence of active autoimmune disease, patients were allowed to use nasal spray, inhalation, or topical corticosteroid drugs, or other corticosteroid drugs with a prednisone equivalent dose ≤10 mg/ day.
18. Receive live vaccination within 4 weeks prior to the initial study administration.
19. Major surgical operations (including primary tumor operations, craniotomy, thoracotomy or laparotomy, etc., excluding vascular access establishment operations) were performed within 4 weeks prior to the first study of drug use.
20. Those who have a history of psychotropic drug abuse and cannot quit or have a history of mental disorders.
21. Pregnant or lactating women.
22. There are other severe, acute, or chronic medical or psychiatric disorders or laboratory abnormalities, as determined by the investigator, that may increase the risks associated with participation in the study or that may interfere with the interpretation of the study findings.
23. Patients who have participated in or are being treated in other clinical trials for any other drug within 28 days prior to the first dose and plan to receive other anticancer therapy or other investigational drug during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities (DLTs) | First Cycle (28 days)
  Number of participants with DLTs during the 28 days following the first administration of FTL008.16

SECONDARY OUTCOMES:
To preliminarily evaluate the anti-tumor activity | Tumor efficacy was evaluated every 8 weeks for the first 56 weeks and every 12 weeks after 56 weeks following calendar days.
  Computed tomography (CT) scans of tumors will be evaluated according to RECIST 1.1 and iRECIST (2017)
Pharmacokinetic (PK) measure: Maximum observed serum concentration (Cmax) | From first dose (Cycle 1 Day 1, each cycle is 28 days) until the last dose (up to 2 years)
  PK samples will be collected at predefined timepoints to determine Cmax.
Pharmacokinetic (PK) measure: Area under the plasma concentration versus time curve (AUC) | From first dose (Cycle 1 Day 1, each cycle is 28 days) until the last dose (up to 2 years)
  PK samples will be collected at predefined timepoints to determine AUC.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Shoubin Wen, MD, Study Director — Sound Biopharmaceuticals Ltd.
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No